CLINICAL TRIAL: NCT00604903
Title: Remon CHF Medical Device Clinical Investigation PAPIRUS II: Monitoring Pulmonary Artery Pressure by Implantable Device Responding to Ultrasonic Signal
Brief Title: Monitoring Pulmonary Artery Pressure by Implantable Device Responding to Ultrasonic Signal
Acronym: PAPIRUSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PAPIRUS II
Record Dates: First submitted 2008-01-04; First posted 2008-01-30 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2012-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients implanted with Pressure Sensor (Experimental): Implant of Pressure sensor. These are patients, who were implanted with the Remon CHF Implantable Pressure Sensor utilizing the corresponding delivering system.
  Interventions: Device: Implant of Pressure sensor.

INTERVENTIONS:
Device: Implant of Pressure sensor. — Implant of an Remon ImPressure implantable pulmonary artery pressure sensor utilizing the corresponding delivering system.

SUMMARY:
The purpose of this study is to evaluate and document appropriate clinical safety and performance of the Remon CHF Implantable Pressure Sensor including the corresponding delivery system, the Remon CHF Home Unit, the Remon CHF Clinic System devices and associated application software. It is a small clinical trial to determine the feasibility of the device. The primary outcome measure relates to feasibility and not to health outcomes.

DETAILED DESCRIPTION:
This study was a prospective feasibility, non-randomised, singlearm, multi-centre, interventional clinical investigation performed at 4 international sites. Patients were implanted with the Remon CHF Implantable Pressure Sensor utilizing the corresponding delivering system. Measurements were taken with the Remon CHF Home Unit and the Remon CHF Clinic System. Follow-up visits took place at one, three and six months after implant.

Per protocol, a minimum of 30 patients was required to demonstrate safety of the device.

The study was conducted in accordance with ISO 14155:2003 (parts I and II), the Declaration of Helsinki and all applicable local and national regulations in the countries of submission.

ELIGIBILITY:
Inclusion Criteria:

* Patients who exhibit signs and symptoms of NYHA Class III or IV heart failure.
* Patients who are able to visit the clinic frequently during the 6 months following implantation.
* Patients who are willing and able to perform all follow-up procedures.

Exclusion Criteria:

1. Patients under the age of 18
2. Pregnant women or women that plan to get pregnant during the study.
3. Patients with, tricuspid or pulmonic stenosis, pulmonary stents, right sided mechanical heart valves
4. Contraindication to antiplatelet therapy (aspirin and clopidogrel)
5. Patients suffering from active infection (on antibiotic therapy)
6. Known intracardiac mass (right atrial or right ventricular)
7. Patients who have been implanted with a VAD
8. Patients who are candidates for listing for heart transplantation if it is deemed that they have a possibility of receiving a heart within the next 6 months
9. Patients that have lead implanted at the heart right side of the heart within the last 6 months
10. Patients with any terminal illness, or with a life expectancy of less than 6 months
11. Patients that are unable to lie flat for the duration of the procedure
12. Patients that are unable to operate the home unit (due to physical or mental constrain)
13. Patients after pneumonectomy
14. Patients treated with oral anticoagulants INR > 1.5 prior to catheterization
15. Patients with severe chronic renal failure (creatinine > 2.5 mg/dl)
16. Patients suffered from acute myocardial infarction within the three months prior the study
17. Patients that underwent open heart surgery within 4 weeks prior the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-08-23 (Actual); Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Serious adverse events related to implantation or the device | 6
  Primary Device Safety Objective: Serious Adverse Device Effects rate during 6 months following implantation (device or delivery system related) and Implantation related Serious Adverse Events rate during 6 months following implantation

SECONDARY OUTCOMES:
Device accuracy | 6 months
  Compare accuracy of Remon Pressure Sensor with Millar catheter (invasive way of measuring pulmonary artery pressure).
  Secondary end points included accuracy of the measured PA pressure, functionality of the system and evaluation of pressure readings at different postures.

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, M.D., Principal Investigator — CardioVascular Center Frankfurt, Seckbacher

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoppe UC, Vanderheyden M, Sievert H, Brandt MC, Tobar R, Wijns W, Rozenman Y. Chronic monitoring of pulmonary artery pressure in patients with severe heart failure: multicentre experience of the monitoring Pulmonary Artery Pressure by Implantable device Responding to Ultrasonic Signal (PAPIRUS) II study. Heart. 2009 Jul;95(13):1091-7. doi: 10.1136/hrt.2008.153486. Epub 2009 Feb 5. PMID 19196733